CLINICAL TRIAL: NCT03081286
Title: Treatment of Postmastectomy Pain Syndrome With Fat Grafting: A Double-blinded Randomized Controlled Trial
Brief Title: Treatment of Postmastectomy Pain Syndrome With Fat Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sollie, Doctor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20160185
Record Dates: First submitted 2017-03-02; First posted 2017-03-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Post-Mastectomy Chronic Pain Syndrome (Disorder)
MeSH Terms: interventions — Lipectomy; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: During general anesthesia, patients are randomized to either fat grafting or sham grafting with only saline. All patients undergo the same liposuction. Participants are blinded, care providers postoperatively are blinded. The surgeon performing the procedure is not blinded. The outcome assessors 3 and 6 months postoperatively are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat grafting (Experimental): Following liposuction the fat is decanted and used for fat grafting to the area of pain after breast cancer surgery.
  Interventions: Procedure: Liposuction; Procedure: Fat graft
- Sham grafting (Sham Comparator): Following liposuction the fat is discarded. Instead approximately 50mL of saline is used instead of fat and injected into the area of pain after breast cancer surgery.
  Interventions: Procedure: Liposuction; Procedure: Sham graft (saline injection)

INTERVENTIONS:
Procedure: Liposuction — Liposuction is performed on the abdomen or thighs as determined before randomization by the surgeon.
Procedure: Fat graft — The harvested lipoaspirate is injected at the site of pain.
  Other Names: lipotransfer
  Arms: Fat grafting
Procedure: Sham graft (saline injection) — Saline will be injected at the site of pain instead of fat
  Arms: Sham grafting

SUMMARY:
This study evaluates the possible beneficial effect of fat grafting for post mastectomy pain syndrome. Half of patients will receive fat grafting and the other half of patients will receive sham.

DETAILED DESCRIPTION:
Several studies have suggested that fat grafting can alleviate pain in post mastectomy pain syndrome. These studies however have either been in the form of case series or unblinded studies with great risk of bias.

It is believed that fat grafting with its content of adipose-derived stem cells can modulate the scar tissue upon grafting and hereby decrease pain.

In this study patients will be randomized to either fat grafting or a sham procedure where they undergo the same liposuction but no fat grafting, only injection of saline instead of fat.

ELIGIBILITY:
Inclusion Criteria:

* Treated for breast cancer
* Pain in the breast cancer treated area on the breast or axilla.
* Pain present at least 4 days a week with an intensity above 3 on VAS.
* Duration longer than 3 months
* Recurrence free for minimum 6 months
* Understand the nature of the study and can give informed consent

Exclusion Criteria:

* Psychiatric condition that can affect participation.
* Recurrence of breast cancer at any time.
* Other indication for fat grafting other than pain treatment.
* Breast reconstruction with flap

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Pain on visual analog scale (VAS) 0-10 | 6 months
  Pain on visual analog scale (VAS) 0-10

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | 3 and 6 months
  Questionnaire
Use of pain medication | 3 and 6 months
  pain medication used is registered on questionnaire
Pain on visual analog scale (VAS) 0-10 | 3 months
  Pain on visual analog scale (VAS) 0-10

OTHER OUTCOMES:
Complications | 3 months
  Any complications following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD PhD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No